CLINICAL TRIAL: NCT05379179
Title: Pilot Study: Ketamine for Acute Pain After Rattlesnake Envenomation
Brief Title: Ketamine Pilot Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: After 20 months of active enrollment and a lack of qualified/interested subjects, the Investigator, Meghan Spyres, MD, decided to terminate recruitment before meeting the stated enrollment objectives.
Sponsor: Meghan Spyres (Other)
Responsible Party: Sponsor-Investigator, Meghan Spyres, Associate Professor, Emergency Medicine, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000919
Record Dates: First submitted 2022-04-15; First posted 2022-05-18 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Rattlesnake Envenomation
Keywords: Acute pain after rattlesnake bite; Rattlesnake envenomation; low dose ketamine; pain dose ketamine
MeSH Terms: interventions — Ketamine; Fentanyl

STUDY DESIGN:
Intervention Model Description: Following enrollment, subject will be randomly assigned to receive either ketamine, or fentanyl. A randomization masterlist has been developed that will be used to assign drug. Subjects will be assigned in sequential order. Each block will alternate between each drug. Subjects will have 50/50 chance of being assigned to ketamine or fentanyl.
Who Masked: Participant
Masking Description: The blinding of the subjects is done by the investigators which is the block randomization; each block will alternate between each drug ketamine or fentanyl. Subject will not be told which pain medication they will receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fentanyl (Active Comparator): Drug administration: A single dose of fentanyl 1mcg/kg IV, maximum 100 mcg, over 15 minutes.
  Time drug given will be documented Data obtained prior to med administration and then following medication administration at intervals of 15, 30, 60 and 120 minutes
  * Record vital signs (HR, B/P, resp rate, O2 sat)
  * Obtain and assess pain response scores
    1. Pain Numerical Rating Score (NRS - 0-10)
    2. Richmond Agitation Sedation Scale (RASS)
    3. Side Effect Rating Scale for Dissociative Anesthesia (SERSDA)
  * Record any airway interventions required? If yes what? new supplemental O2/BVM/intubation, jaw thrust
  * Record any rescue meds, dose and time (Rescue medication - Fentanyl):
  * 1 mcg/kg IV fentanyl (0.5 mcg/kg if age >55 yrs)
  * Defined as rescue if given <30 min post study intervention for pain score >5 or patient requesting additional medication.
  * Patient pain satisfaction score at discharge
  Interventions: Drug: Fentanyl
- Ketamine (Experimental): Drug administration: A single dose of ketamine 0.3 mg/kg IV over 15 minutes. Time drug given will be documented Data obtained prior to med administration and then following medication administration at intervals of 15, 30, 60 and 120 minutes
  * Record vital signs (HR, B/P, resp rate, O2 sat)
  * Obtain and assess pain response scores
    1. Pain Numerical Rating Score (NRS - 0-10)
    2. Richmond Agitation Sedation Scale (RASS)
    3. Side Effect Rating Scale for Dissociative Anesthesia (SERSDA)
  * Record any airway interventions required? If yes what? new supplemental O2/BVM/intubation, jaw thrust
  * Record any rescue meds, dose and time (Rescue medication - Fentanyl):
  * 1 mcg/kg IV fentanyl (0.5 mcg/kg if age >55 yrs)
  * Defined as rescue if given <30 min post study intervention for pain score >5 or patient requesting additional medication.
  * Patient pain satisfaction score at discharge
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — This study will compare patient-reported pain scores after receiving either ketamine or fentanyl for the treatment of acute pain due to a rattlesnake bite.
  Arms: Ketamine
Drug: Fentanyl — This study will compare patient-reported pain scores after receiving either ketamine or fentanyl for the treatment of acute pain due to a rattlesnake bite.
  Arms: Fentanyl

SUMMARY:
This is a pilot study to evaluate pain responses from two different approved medications (ketamine and fentanyl) in the treatment of pain after rattlesnake envenomation (RSE). Both medications are currently used in standard practice to treat both acute and chronic pain and are options for pain management after RSE. Multiple studies exist showing ketamine to be both safe and effective for the treatment of acute pain, and to be as good as or better than opioids for this indication. The specific comparison of ketamine to fentanyl, however, has never been studied for the treatment of acute pain after rattlesnake envenomation in the United States. The investigators plan to measure pain scores after a single dose of ketamine or fentanyl in patients shortly after being envenomated, followed by continued treatment of pain guided by the treating doctor. There will be no restrictions on additional pain medications given and no other changes to the treatment of these patients during their hospitalization. This research is important because pain after RSE can be difficult to control and may require frequent, high doses of opioids for several days. An effective non-opioid medication would be helpful both to better-control pain and to reduce exposure to opioids in this patient population. This study will compare patient-reported pain scores after receiving a single dose of ketamine or fentanyl in patients with rattlesnake bites who have been admitted to the toxicology service at Banner - University Medical Center Phoenix (BUMCP).

DETAILED DESCRIPTION:
Multiple studies have shown ketamine to be safe and effective agent for acute pain syndromes. RSEs classically result in severe pain that can be difficult to control, despite use of opioids, non-opioid analgesics, and positioning techniques, including splinting and elevation. Furthermore, the ongoing opioid epidemic pushes clinicians to explore non-opioid agents to avoid unnecessary exposure of patients to these high-risk medications. At least one small study has shown ketamine to be safe in rattlesnake envenomated patients.

ELIGIBILITY:
Inclusion Criteria:

* Ages ≥ 18 years.
* Able to speak and understand English.
* RSE requiring IV pain medication for NRS pain score > 5.
* No allergy to ketamine or fentanyl.
* Ability to provide informed consent.
* ≤ 24 hours from envenomation.

Exclusion Criteria:

* Pregnant or lactating.
* Prisoners.
* Refugees.
* History of schizophrenia.
* Clinically intoxicated.
* On buprenorphine therapy.
* History of uncontrolled hypertension
* Increased intracranial pressure
* Systemic envenomation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-08-27 (Actual); Study Completion 2022-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Spyres, MD, Principal Investigator — University of Arizona
Locations (1):
- Banner - University Medical Center, Phoenix campus, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Karlow N, Schlaepfer CH, Stoll CRT, Doering M, Carpenter CR, Colditz GA, Motov S, Miller J, Schwarz ES. A Systematic Review and Meta-analysis of Ketamine as an Alternative to Opioids for Acute Pain in the Emergency Department. Acad Emerg Med. 2018 Oct;25(10):1086-1097. doi: 10.1111/acem.13502. Epub 2018 Jul 17. PMID 30019434
- [Background] Brandehoff N, Benjamin JM, Balde C, Chippaux JP. Ketamine for pain control of snake envenomation in Guinea: A case series. Toxicon. 2020 Nov;187:82-85. doi: 10.1016/j.toxicon.2020.08.020. Epub 2020 Sep 3. PMID 32891662
- [Background] Balzer N, McLeod SL, Walsh C, Grewal K. Low-dose Ketamine For Acute Pain Control in the Emergency Department: A Systematic Review and Meta-analysis. Acad Emerg Med. 2021 Apr;28(4):444-454. doi: 10.1111/acem.14159. Epub 2021 Jan 2. PMID 33098707
- [Background] Andolfatto G, Willman E, Joo D, Miller P, Wong WB, Koehn M, Dobson R, Angus E, Moadebi S. Intranasal ketamine for analgesia in the emergency department: a prospective observational series. Acad Emerg Med. 2013 Oct;20(10):1050-4. doi: 10.1111/acem.12229. PMID 24127709
- [Background] Gallagher EJ, Liebman M, Bijur PE. Prospective validation of clinically important changes in pain severity measured on a visual analog scale. Ann Emerg Med. 2001 Dec;38(6):633-8. doi: 10.1067/mem.2001.118863. PMID 11719741

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from patients hospitalized with rattlesnake bites at Banner University Medical Center between 05/2022 and 01/2024. The first participant was enrolled on 06/20/2022, and the last was enrolled in 08/2022.
Pre-assignment Details: Of the 3 enrolled participants, 3 met inclusion criteria and were randomized.
Groups:
- Fentanyl: Drug administration: A single dose of fentanyl 1mcg/kg IV, maximum 100 mcg, over 15 minutes.
  Time drug given will be documented Data obtained prior to med administration and then following medication administration at intervals of 15, 30, 60 and 120 minutes
  * Record vital signs (HR, B/P, resp rate, O2 sat)
  * Obtain and assess pain response scores
    1. Pain Numerical Rating Score (NRS - 0-10)
    2. Richmond Agitation Sedation Scale (RASS)
    3. Side Effect Rating Scale for Dissociative Anesthesia (SERSDA)
  * Record any airway interventions required? If yes what? new supplemental O2/BVM/intubation, jaw thrust
  * Record any rescue meds, dose and time (Rescue medication - Fentanyl):
  * 1 mcg/kg IV fentanyl (0.5 mcg/kg if age >55 yrs)
  * Defined as rescue if given <30 min post study intervention for pain score >5 or patient requesting additional medication.
  * Patient pain satisfaction score at discharge
  Fentanyl: This study will compare patient-reported pain scores after receiving either ketamine or fentanyl for the treatment of acute pain due to a rattlesnake bite.
- Ketamine: Drug administration: A single dose of ketamine 0.3 mg/kg IV over 15 minutes. Time drug given will be documented Data obtained prior to med administration and then following medication administration at intervals of 15, 30, 60 and 120 minutes
  * Record vital signs (HR, B/P, resp rate, O2 sat)
  * Obtain and assess pain response scores
    1. Pain Numerical Rating Score (NRS - 0-10)
    2. Richmond Agitation Sedation Scale (RASS)
    3. Side Effect Rating Scale for Dissociative Anesthesia (SERSDA)
  * Record any airway interventions required? If yes what? new supplemental O2/BVM/intubation, jaw thrust
  * Record any rescue meds, dose and time (Rescue medication - Fentanyl):
  * 1 mcg/kg IV fentanyl (0.5 mcg/kg if age >55 yrs)
  * Defined as rescue if given <30 min post study intervention for pain score >5 or patient requesting additional medication.
  * Patient pain satisfaction score at discharge
  Ketamine: This study will compare patient-reported pain scores after receiving either ketamine or fentanyl for the treatment of acute pain due to a rattlesnake bite.
Period: Overall Study
Arm/Group | Fentanyl | Ketamine
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fentanyl | Ketamine | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Assessment Post Medication
Description: Pain will be assessed using a numerical rating scale (0-10, with 0 being no pain and 10 being the worst pain) at 30, 60, and 120 minutes after medication administration.
Time Frame: 30-120 minutes after drug administration
Population: Note there was only 1 patient in the Ketamine group thus medians represent this single patient value, no range calculated.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Fentanyl | Ketamine
Number analyzed (Participants) | 2 | 1
units on a scale
  30 minutes | 1 [1 to 1] | 10
  60 minutes | 1.5 [1.25 to 1.75] | 5
  120 minutes | 1.5 [1.25 to 1.75] | 10

2. Secondary Outcome: Adverse Events
Description: A subjects chart will be reviewed to determine whether rescue medication was needed or if there were any adverse medications effects
Time Frame: During hospitalization, up to 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Fentanyl | Ketamine
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: During hospitalization, up to 120 minutes.
Description: A subjects chart will be reviewed to determine whether rescue medication was needed or if there were any adverse medications effects.
Arm/Group | Fentanyl | Ketamine
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

LIMITATIONS AND CAVEATS:
Significant limitations were not reaching the target number of patients, extremely low enrollment resulted in termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT05379179/Prot_SAP_000.pdf